CLINICAL TRIAL: NCT03068624
Title: Phase Ib Study of Cellular Adoptive Immunotherapy Using Autologous Cd8+ Antigen-Specific T Cells and Anti-Ctla4 for Patients With Metastatic Uveal Melanoma
Brief Title: Autologous CD8+ SLC45A2-Specific T Lymphocytes With Cyclophosphamide, Aldesleukin, and Ipilimumab in Treating Patients With Metastatic Uveal Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0414; NCI-2018-01291 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0414 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-02-24; First posted 2017-03-03 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Malignant Neoplasm in the Liver; Metastatic Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — aldesleukin; Cyclophosphamide; Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cyclophosphamide, T-cells, aldesleukin, ipilimumab) (Experimental): PREPARATIVE REGIMEN: Patients receive cyclophosphamide IV over 30-60 minutes on day -2.
  T-CELL INFUSION: Patients receive autologous CD8+ SLC45A2-specific T lymphocytes via hepatic arterial infusion via central catheter over 60 minutes on day 0. Within 6 hours of T-cell infusion, patients also receive aldesleukin BID SC for 14 days in the absence of disease progression or unacceptable toxicity.
  POST T-CELL INFUSION: Patients receive ipilimumab IV over 90 minutes on days 1, 22, 43, and 64 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Aldesleukin; Biological: Autologous CD8+ SLC45A2-specific T Lymphocytes; Drug: Cyclophosphamide; Biological: Ipilimumab

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: Autologous CD8+ SLC45A2-specific T Lymphocytes — Given via hepatic arterial infusion via central catheter
  Other Names: Autologous SLC45A2-specific CTLs; Autologous SLC45A2-specific Cytotoxic T Lymphocytes
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy

SUMMARY:
This phase Ib trial studies the side effects and best dose of autologous CD8 positive (+) SLC45A2-specific T lymphocytes when given together with cyclophosphamide, aldesleukin, and ipilimumab, and to see how well they work in treating patients with uveal melanoma that has spread to other places in the body (metastatic). To make specialized CD8+ T cells, researchers separate out T cells collected from patients' blood and treat them so they are able to target melanoma cells. The blood cells are then given back to the patients. This is known as "adoptive T cell transfer" or "adoptive T cell therapy." Drugs used in chemotherapy, such as cyclophosphamide, may work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Biological therapies, such as aldesleukin, use substances made from living organisms that may stimulate the immune system in different ways and stop tumor cells from growing. Immunotherapy with monoclonal antibodies, such as ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving autologous CD8+ SLC45A2-specific T lymphocytes together with cyclophosphamide, aldesleukin, and ipilimumab may work better in treating patients with metastatic uveal melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) of adoptively transferred SLC45A2-specific cytotoxic T-lymphocytes (CTL) for the treatment of patients with metastatic uveal melanoma.

SECONDARY OBJECTIVES:

I. To establish the anti-tumor efficacy as measured by immune-related response criteria (irRC) and duration of response in metastatic uveal melanoma patients receiving autologous CD8+ T cells against SLC45A2.

II. To assess the safety and tolerability of adoptively transferred SLC45A2-specific CTL in combination with immune checkpoint blockade in metastatic uveal melanoma patients.

III. To quantify in vivo numeric and functional persistence of transferred CTL, and development of antigen spreading in metastatic uveal melanoma patients.

IV. To assess overall survival and progression-free survival in metastatic uveal melanoma patients.

OUTLINE: This is a dose escalation study of autologous CD8+ SLC45A2-specific T lymphocytes.

PREPARATIVE REGIMEN: Patients receive cyclophosphamide intravenously (IV) over 30-60 minutes on day -2.

T-CELL INFUSION: Patients receive autologous CD8+ SLC45A2-specific T lymphocytes via hepatic arterial infusion via central catheter over 60 minutes on day 0. Within 6 hours of T-cell infusion, patients also receive aldesleukin twice daily (BID) subcutaneously (SC) for 14 days in the absence of disease progression or unacceptable toxicity.

POST T-CELL INFUSION: Patients receive ipilimumab IV over 90 minutes on days 1, 22, 43, and 64 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at days 84 and 168, and then every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* PHERESIS (TURNSTILE 1): Histopathologic documentation of melanoma concurrent with the diagnosis of metastatic disease or high-risk primary uveal melanoma defined as a recurrence score of > 50% in 5 years. A diagnosis of uveal melanoma can be made clinically without primary tissue evaluation, based on history and records. A prior history of brachytherapy to the eye is sufficient clinical support for a diagnosis of uveal melanoma.
* PHERESIS (TURNSTILE 1): Hematocrit (HCT) >= 24% or hemoglobin (HB) >= 8 g/dL.
* PHERESIS (TURNSTILE 1): Platelets > 50,000.
* PHERESIS (TURNSTILE 1): Expression of human leukocyte antigen (HLA)-A:0201 or HLA-A:2402.
* PHERESIS (TURNSTILE 1): Eastern Cooperative Oncology Group (ECOG)/ Zubrod performance status of 0-1.
* PHERESIS (TURNSTILE 1): Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized. Suggested precautions should be used to minimize the risk or pregnancy for at least 1 month before start of therapy, and while women are on study for up to 3 months after completion of the study. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal.
* PHERESIS (TURNSTILE 1): Male patients must be willing and able to use an acceptable method of birth control, during and for at least 3 months after completion of the study, if their sexual partners are WOCBP.
* PHERESIS (TURNSTILE 1): Willing and able to give informed consent.
* PHERESIS (TURNSTILE 1): Toxicity related to prior therapy must either have returned to =< grade 1, baseline, or been deemed irreversible. Certain non-serious exceptions include alopecia, hypothyroidism, neuropathy, nausea, adrenocortical deficiency requiring physiologic replacement dose of steroids, and other conditions noted and approved by the principal investigator (PI).
* T CELL INFUSION (INCLUDES CYCLOPHOSPHAMIDE, T CELL, ANTI-CTLA4 INFUSIONS AND SC IL-2) (TURNSTILE 2): ECOG/Zubrod performance status of 0-1 (evaluate at least 1 week before T cell infusion).
* T CELL INFUSION (INCLUDES CYCLOPHOSPHAMIDE, T CELL, ANTI-CTLA4 INFUSIONS AND SC IL-2) (TURNSTILE 2): Bi-dimensionally measurable disease by palpation on clinical exam, or radiographic imaging per irRC (evaluate at least 1 week before T cell infusion).
* T CELL INFUSION (INCLUDES CYCLOPHOSPHAMIDE, T CELL, ANTI-CTLA4 INFUSIONS AND SC IL-2) (TURNSTILE 2): At least 4 weeks must have elapsed since the last chemotherapy, targeted therapy, immunotherapy, radiotherapy, liver-directed therapy, or major surgery. At least 6 weeks for nitrosoureas, mitomycin C and liposomal doxorubicin. If started before T-cell administration, ipilimumab infusions must be least 21 days apart (evaluate at least 1 week before T cell infusion).
* T CELL INFUSION (INCLUDES CYCLOPHOSPHAMIDE, T CELL, ANTI-CTLA4 INFUSIONS AND SC IL-2) (TURNSTILE 2): For the ipilimumab cohort only: Toxicity related to prior therapy must either have returned to =< grade 1, baseline, or been deemed irreversible. Certain non-serious exceptions include alopecia, hypothyroidism, neuropathy, nausea, adrenocortical deficiency requiring physiologic replacement dose of steroids, and other conditions noted and approved by the PI (evaluate at least 1 week before T cell infusion).
* T CELL INFUSION (INCLUDES CYCLOPHOSPHAMIDE, T CELL, ANTI-CTLA4 INFUSIONS AND SC IL-2) (TURNSTILE 2): Patients must have liver metastasis (evaluate at least 1 week before T cell infusion).
* T CELL INFUSION (INCLUDES CYCLOPHOSPHAMIDE, T CELL, ANTI-CTLA4 INFUSIONS AND SC IL-2) (TURNSTILE 2): Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 3 months after completion of study (evaluate at least 1 week before T cell infusion).
* T CELL INFUSION (INCLUDES CYCLOPHOSPHAMIDE, T CELL, ANTI-CTLA4 INFUSIONS AND SC IL-2) (TURNSTILE 2): Willing and able to give informed consent (evaluate at least 1 week before T cell infusion).

Exclusion Criteria:

* PHERESIS: Secondary malignancy is allowed providing it does not require concurrent therapy.
* PHERESIS: Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception. Women of childbearing potential with a positive pregnancy test within 3 days prior to pheresis.
* PHERESIS: Significant cardiovascular abnormalities as defined by any one of the following:

  * Congestive heart failure
  * Clinically significant hypotension
  * Symptoms of coronary artery disease (angina, dyspnea)
  * Presence of cardiac arrhythmias on electrocardiogram (EKG) requiring drug therapy
* PHERESIS: Autoimmune disease: Patients with a history of inflammatory bowel disease are excluded from this study, as are patients with a history of autoimmune disease (e.g. systemic lupus erythematosus, vasculitis, infiltrating lung disease) whose possible progression during treatment would be considered by the investigator to be unacceptable. Acceptable exclusions include: Hashimoto's thyroiditis, type 1 diabetes mellitus, and other localized or inactive conditions with approval of the PI.
* PHERESIS: Any underlying medical or psychiatric condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea.
* PHERESIS: Positive screening tests for human immunodeficiency virus (HIV), hepatitis B virus (Hep B), and hepatitis C virus (Hep C). If positive results are not indicative of true active or chronic infection, the patient can be treated.
* PHERESIS: Participation in any other immunotherapy treatment, that in the opinion of the principal investigator would be unsafe to receive further checkpoint blockade immunotherapy
* White blood cell (WBC) =< 2000/uL (prior to cyclophosphamide and T cell infusions).
* Hct =< 24% or Hb =< 8 g/dL (prior to cyclophosphamide and T cell infusions).
* Absolute neutrophil count (ANC) =< 1000 (prior to cyclophosphamide and T cell infusions).
* Platelets =< 50,000 (prior to cyclophosphamide and T cell infusions).
* Creatinine >= 3.0 x upper limit of normal (ULN) (prior to cyclophosphamide and T cell infusions).
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >= 5 x ULN (since all patients will have liver metastasis) (prior to cyclophosphamide and T cell infusions).
* Bilirubin >= 3 x ULN (prior to cyclophosphamide and T cell infusions).
* Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception. Women of childbearing potential with a positive pregnancy test within 3 days prior to entry.
* Clinically significant pulmonary dysfunction, as determined by medical history and physical exam. Patients so identified will undergo pulmonary functions testing and those with forced expiratory volume in one second (FEV1) < 2.0 L or diffusing capacity of the lung for carbon monoxide (DLCO) (corrected [corr] for hemoglobin [Hgb]) < 50% will be excluded.
* Steroids (at prednisone equivalent doses > 10 mg) are not permitted 3 days prior to T cell infusion and concurrently during therapy. Exceptions include use of systemic prednisone equivalent doses =< 10 mg/ day, topical steroids or physiologic replacement dose of steroids for adrenocortical deficiency.
* Any non-oncology vaccine therapy used for the prevention of infectious disease within 1 month before or after any ipilimumab dose.
* Patients may not be on any other treatments for their cancer aside from those included in the protocol. Patients may not undergo another form of treatment concurrently with this study. Oncology supportive treatments such as growth factors, bone modifying agents, pain or nausea management are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 6 weeks
  As determined by dose limiting toxicity (DLT). MTD defined at the highest dose at which no more than 1 in 6 patients has experienced DLT.

SECONDARY OUTCOMES:
Overall response rate | Up to 5 years
  As measured by immune-related response criteria. Overall response will be monitored simultaneously using the Bayesian approach of Thall, Simon, Estey and the extension by Thall and Sung. Logistic regression will be used to assess the impact of patient characteristics on the overall response rate.
Duration of clinical response (DOR) | From the start of study treatment up to 5 years
  DOR will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups of patients will be made using the log-rank test. Cox (proportional hazards) regression will be used to evaluate multivariable predictive models of time-to-event outcomes. Continuous variables (e.g., age, etc.) will be summarized using the mean (standard deviation) or median (range). Frequency tables will be used to summarize categorical variables.
Persistence of in vivo T cells and non-target antigen recognition | From the start of study treatment up to 5 years
  Continuous variables (e.g., age, etc.) will be summarized using the mean (standard deviation) or median (range). Frequency tables will be used to summarize categorical variables. The distribution of time-to-event endpoints will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups of patients will be made using the log-rank test. Cox proportional hazards) regression will be used to evaluate multivariable predictive models of time-to-event outcomes.
Overall survival (OS) | From the start of study treatment up to 5 years
  OS will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups of patients will be made using the log-rank test. Cox (proportional hazards) regression will be used to evaluate multivariable predictive models of time-to-event outcomes. Continuous variables (e.g., age, etc.) will be summarized using the mean (standard deviation) or median (range). Frequency tables will be used to summarize categorical variables.
Progression-free survival (PFS) | From the start of study treatment up to 5 years
  PFS will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups of patients will be made using the log-rank test. Cox (proportional hazards) regression will be used to evaluate multivariable predictive models of time-to-event outcomes. Continuous variables (e.g., age, etc.) will be summarized using the mean (standard deviation) or median (range). Frequency tables will be used to summarize categorical variables.
Time to response | From the start of study treatment up to 5 years
  Continuous variables (e.g., age, etc.) will be summarized using the mean (standard deviation) or median (range). Frequency tables will be used to summarize categorical variables. The distribution of time-to-event endpoints will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups of patients will be made using the log-rank test. Cox proportional hazards) regression will be used to evaluate multivariable predictive models of time-to-event outcomes.
Incidence of toxicity | Up to 5 years
  Toxicity will be monitored simultaneously using the Bayesian approach of Thall, Simon, Estey and the extension by Thall and Sung. An Efficacy/ Summary will be submitted to the Investigational New Drug (IND) Office Medical Monitor after every six evaluable patients complete 12 weeks of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sapna P Patel, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org